CLINICAL TRIAL: NCT04445467
Title: An Adaptive Randomised Placebo Controlled Phase II Trial of Antivirals for COVID-19 Infection
Brief Title: An Adaptive Clinical Trial of Antivirals for COVID-19 Infection
Acronym: VIRCO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 66223
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: COVID
MeSH Terms: interventions — favipiravir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Favipiravir (Experimental): 1800 mg Favipiravir twice daily on Day 1 followed by 800 mg Favipiravir twice daily for the next 13 days.
  Interventions: Drug: Favipiravir
- Placebo (Placebo Comparator): Matched Placebo
  Interventions: Drug: Favipiravir

INTERVENTIONS:
Drug: Favipiravir — Favipiravir

SUMMARY:
This is a randomised placebo controlled phase II trial to examine the efficacy of antivirals to treat COVID-19 infection compared to placebo for virological cure and improved clinical outcomes. Individuals will be randomised to the candidate antiviral which in the first instance is Favipiravir or matched placebo and randomisation will be stratified according to whether the participant requires hospitalisation or not. This treatment will be given in addition to the usual standard of care in the participating hospital.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent by the participant or authorized representative
* Age ≥18 years
* Confirmed SARS-CoV-2 by nucleic acid testing in the past 5 days
* COVID-19 related symptom initiation within 5 days
* Female patients of childbearing potential must have a negative pregnancy test at Screening. Female patients of childbearing potential and fertile male patients who are sexually active with a female of childbearing potential must use highly effective methods of contraception throughout the study and for 1 week following the last dose of study treatment.

Exclusion Criteria:

* Known allergy to the study medication
* Is on another antiviral for the treatment of COVID-19
* Pregnancy
* Patients with severe hepatic dysfunction equivalent to Grade C in the Child-Pugh classification
* Patients with renal impairment requiring dialysis
* Is deemed by the Investigator to be ineligible for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Time to virological cure | 14 days
  Time to 2 successive throat (or combined nose/throat) swabs negative for SARS-CoV-2 by nucleic acid testing

SECONDARY OUTCOMES:
Safety | 28 days
  All adverse events definitely, probably or possibly related to study treatment.
Clinical improvement | 28 days
  Time from randomization to an improvement of two points (from the status at randomization) on the 7-point ordinal scale
Clinical symptoms | 28 days
  Time from randomization to resolution of clinical symptoms (fever, cough, shortness of breath, cough). Resolution defined as the start of the first 24 hour period when all symptoms are rated as mild or absent and remained this way for 24 hours
Biomarkers | 28 days
  Biomarkers taken as part of routine care including total lymphocyte count, CRP, Ferritin and LDH.

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] McMahon JH, Lau JSY, Roney J, Rogers BA, Trubiano J, Sasadeusz J, Molton JS, Gardiner B, Lee SJ, Hoy JF, Cheng A, Peleg AY. An adaptive randomised placebo controlled phase II trial of antivirals for COVID-19 infection (VIRCO): A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Oct 13;21(1):847. doi: 10.1186/s13063-020-04766-5. PMID 33050947